CLINICAL TRIAL: NCT01504165
Title: A Phase I, Open-label, Parallel-group, Mono-center Trial to Investigate the Pharmacokinetics of a Single Intravenous Dose of Cilengitide in Subjects With Mild, Moderate or Severe Renal Impairment Compared to Subjects With Normal Renal Function
Brief Title: Pharmacokinetics in Subjects With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: EMR062041_016; 2011-002389-19 (EudraCT Number)
Record Dates: First submitted 2012-01-03; First posted 2012-01-05 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Renal Impairment
Keywords: Renal impairment; Pharmacokinetic; cilengitide; subjects with mild; moderate or severe renal impairment compared to subjects with normal renal function
MeSH Terms: conditions — Renal Insufficiency; Lymphoma, Follicular | interventions — Cilengitide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group 1 (Experimental): Healthy volunteers: matched subjects with normal renal function
  Interventions: Drug: cilengitide 2000mg
- Group 2 (Experimental): Mild renal impaired subjects
  Interventions: Drug: cilengitide 2000mg
- Group 3 (Experimental): Moderate renal impaired subjects
  Interventions: Drug: cilengitide 2000mg
- Group 4a (Experimental): First group of Severe renal impaired subjects
  Interventions: Drug: cilengitide 1000mg
- Group 4b (Experimental): Second group of severe renal impaired subjects
  Interventions: Drug: cilengitide > 1000mg and up to 2000mg

INTERVENTIONS:
Drug: cilengitide 2000mg — A single dose of cilengitide 2000mg (250mL) will be administered as 1-hour i.v. infusion on Day 1
  Arms: Group 1
Drug: cilengitide 2000mg — A single dose of cilengitide 2000mg (250mL) will be administered as 1-hour i.v. infusion on Day 1
  Arms: Group 2
Drug: cilengitide 2000mg — A single dose of cilengitide 2000mg (250mL) will be administered as 1-hour i.v. infusion on Day 1
  Arms: Group 3
Drug: cilengitide 1000mg — A single dose of cilengitide 1000mg (125mL) will be administered as 1-hour i.v. infusion on Day 1
  Arms: Group 4a
Drug: cilengitide > 1000mg and up to 2000mg — A single dose of cilengitide > 1000mg and up to 2000mg will be administered as 1-hour i.v. infusion on Day 1 if applicable, based on Safety Monitoring Committee decision
  Arms: Group 4b

SUMMARY:
This is an open-label, non-randomized, parallel-group, mono-center, single intravenous dose, Phase I trial to investigate the Pharmacokinetic (PK) and safety of cilengitide in subjects with different grades of renal impairment as compared to subjects with normal renal function.

DETAILED DESCRIPTION:
Subjects with impaired renal function will be screened and will be stratified by their estimated glomerular filtration rate (GFR) according to the Modification of Diet in Renal Disease (MDRD) equation and assigned to one of the stratification groups defined below:

Group Number/Renal function/Creatinine Clearance (GFR according to MDRD)

1. Normal renal function (≥ 90 mL/min)
2. Mild renal impairment (60 - 89 mL/min)
3. Moderate renal impairment (30 - 59 mL/ min) 4a: Severe renal impairment (< 30 mL/min) - no dialysis required 4b: (if applicable) Severe renal impairment (< 30 mL/min) - no dialysis required

Subjects in Groups 2 and 3 will receive a single dose of 2000mg of cilengitide as 1-hour i.v. infusion. Subjects from group 4a will receive a single dose of 1000mg of cilengitide as 1-hour i.v. infusion . PK samples will be collected and basic PK parameters will be calculated. The safety, tolerability, and PK will be evaluated by the Safety Monitoring Committee (SMC). If the SMC has no concerns, Group 4b will be treated with a higher dose (up to 2000mg) of cilengitide. Then, Group 1 (healthy subjects) will be started after the last subject with renal impairment (in either Group 2, 3, or 4a; or in Group 4b, if applicable) has completed all activities on Day 3. They will also receive a single dose of 2000mg of cilengitide as 1-hour i.v. infusion.

The duration of the trial from the first subject enrolled to the last subject last visit will be approximately 6 months (approximately 8 months, in case Group 4b is included). Each subject will participate in the trial for up to 35 days, including screening and the end of trial examination.

ELIGIBILITY:
Inclusion Criteria:

- Body mass index (BMI): ≥ 18 kg/m² and ≤ 35 kg/m²

For subjects with normal renal function:

* Vital signs (pulse rate and blood pressure) within the normal range or showing no clinically relevant deviation
* Estimated creatinine clearance according to the MDRD equation of ≥ 90 mL/min at Screening

For subjects with impaired renal function:

* Laboratory parameters should be within acceptable range for subjects with renal impairment,
* Vital signs: Pulse rate within the normal range of 45-100 beats/minute in supine position after 5 minutes of rest. Blood pressure diastolic below 100 mmHg, and systolic below 160 mmHg for Groups 1-3 and below 180 mmHg for Group 4a and 4b, in supine position after 5 minutes of rest
* Calculated creatinine clearance according to the MDRD equation of < 90 mL/min at Screening and the possibility of stratification to one of the Groups.

Exclusion Criteria:

* History of malignant disease within the last 5 years or acute malignant disease
* Medical history of wound healing problems and/or any current open wounds
* Current or history of bleeding disorders and/or history of thromboembolic events (considering family history as well); thrombolytics or oral or parenteral anticoagulants within 30 days prior to Day 1
* Electrocardiogram recording (12-lead ECG) with signs of clinically relevant pathology as judged by the Investigator

For subjects with impaired renal function:

* Chronic heart failure non stabilized (New York Heart Association [NYHA] class III and IV)
* Acute renal failure of any etiology (including viral, toxic, or drug induced)
* Requiring dialysis
* History of renal transplantation
* Uncontrolled diabetes mellitus as judged by the Investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of cilengitide in plasma | 48 hours after start of infusion of 1 single dose of cilengitide administered as 1-hour intravenous infusion
  Cmax of cilengitide in plasma after single dose in groups of subjects with different grades of renal function compared to subjects with normal renal function.
Area under the plasma concentration versus time curve (AUC) of cilengitide in plasma | 48 hours after start of infusion of 1 single dose of cilengitide administered as 1-hour intravenous infusion
  AUC of cilengitide in plasma after single dose in groups of subjects with different grades of renal function compared to subjects with normal renal function.

SECONDARY OUTCOMES:
Terminal half life t1/2 of cilengitide | 48 hours after start of infusion of 1 single dose of cilengitide administered as 1-hour intravenous infusion
Plasma clearance of cilengitide (CL) | 48 hours after start of infusion of 1 single dose of cilengitide administered as 1-hour intravenous infusion
Cilengitide volume of distribution (Vz) in plasma | 48 hours after start of infusion of 1 single dose of cilengitide administered as 1-hour intravenous infusion
Absolute and relative amount of cilengitide excreted into urine (Ae0-∞) | 24 hours after start of infusion of 1 single dose of cilengitide administered as 1-hour intravenous infusion
Renal clearance of cilengitide (CLR) | 24 hours after start of infusion of 1 single dose of cilengitide administered as 1-hour intravenous infusion
Plasma-protein-binding: Fraction unbound of cilengitide | 2 hours after start of infusion of 1 single dose of cilengitide administered as 1-hour intravenous infusion

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Becker, MD MSc, Study Director — Merck Serono S.A., Geneva
Locations (2):
- Germany (2):
  - For Research Sites contact Merck KGaA Communication Center in, Darmstadt
  - CRS Clincial Research Services Kiel GmbH, Kiel